CLINICAL TRIAL: NCT05100446
Title: Prospective Randomized Trial: Comparison Between High-dose Amoxicillin Dual Therapy and Pylera Quadruple Therapy in the Treatment of Helicobacter Pylori Infection
Brief Title: Comparison Between High-dose Amoxicillin Dual Therapy and Pylera Quadruple Therapy in the Treatment of Helicobacter Pylori Infection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde do Alto Ave, EPE (Other)
Responsible Party: Principal Investigator, Vitor Bruno Macedo da Silva, Medical Doctor, Unidade Local de Saúde do Alto Ave, EPE
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101/2020
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Helicobacter Pylori Infection; Gastritis; Gastric Cancer
MeSH Terms: conditions — Gastritis; Stomach Neoplasms | interventions — Amoxicillin; Esomeprazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Pylera (r) + esomeprazole 40mg (Active Comparator)
  Interventions: Drug: Pylera; Drug: Esomeprazole 40mg
- Treatment with high-dose amoxicillin + esomeprazole 40mg (Active Comparator)
  Interventions: Drug: Amoxicillin - high dose dual therapy; Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: Amoxicillin - high dose dual therapy — Eradication with Amoxicillin 1000mg + 500 mg + 1000mg + 500mg, for 15 days.
  Arms: Treatment with high-dose amoxicillin + esomeprazole 40mg
Drug: Pylera — Eradication with Pylera, for 10 days.
  Arms: Treatment with Pylera (r) + esomeprazole 40mg
Drug: Esomeprazole 40mg — Esomeprazole 40mg, twice a day.

SUMMARY:
Helicobacter pylori is a pathogenic bacteria transmitted from individual to individual, being scientifically recognized as an agent who causes persistent inflammatory activity on the gastric mucosa. This pathogen represents a Global Health problem, as shown in a systematic review by Hooi et al. Besides regional differences, more that half of the world population is expected to have already been infected by this bacteria.

In Portugal, research studies estimate that more than 80% of the adult population has already contacted with H. pylori.

H. pylori infection is associated with active chronic gastritis in every colonized patient, what may consequently lead to peptic ulcer disease, atrophic gastritis, gastric adenocarcinoma and mucosa-associated lymphoid tissue (MALT) lymphoma.

For that reason, H. pylori infection is considered to be a disease, independently of the presence of gastrointestinal symptoms. Additionally, H. pylori has been classified as a confirmed carcinogen (class I) by the International Agency for Research, being responsible for carcinogenic pathways conducting to both gastric adenocarcinoma and lymphoma. This fact gains a particular relevance taking into account that gastric cancer is one of the most prevalent cancers worldwide. On other hand, more than 75% of the gastric cancers occur following H. pylori infection.

Thus, H. pylori eradication constitutes an essential Public Health measurement, being inclusively considered a cost-effective method to decrease the gastric cancer burden, by promoting pre-malignant lesions regression, such as atrophic gastritis, and by delaying the disease progression in case of intestinal metaplasia or dysplasia.

Maastricht V consensus is a document updated in 2016, including the major recommendations regarding H. pylori diagnosis, follow-up and treatment. It highlights the emergence of antibiotic resistances and how they must influence clinical practice, namely the choice of antibiotic regimens, as successful eradication has become less frequent with more prevalent antibiotic resistances. This is the case of clarithromycin and metronidazol, both currently recommended as first-line options by the Portuguese Society of Gastroenterology. In fact, a systematic review conducted in 2018, aiming to evaluate antibiotic resistances on the Portuguese population observed that clarithromycin, metronidazole and double resistance occurred in 42%, 25% and 20% of the individuals, respectively.

Nowadays, Maastricht V guidelines recommend quadruple regimens containing bismuth, such as Pylera (r), as the first-line option in areas with significant double resistance to metronidazole and clarithromycin. Another option currently being investigated is the double therapy with amoxicillin in high doses and proton pump inhibitor. This has become a particularly attractive alternative due to its efficacy, good tolerability and significantly low resistance (<1%) among the European population.

The aim of this clinical trial is to compare both regimens - pylera (r) and high-dose amoxycillin - in H. pylori eradication, regarding their efficacy, tolerability and side effects, in order to asses viable therapeutic options in a population with progressively increasing resistances to alternative regimens currently recommended.

ELIGIBILITY:
Inclusion Criteria:

* Documented Helicobacter pylori infection
* Age equal or greater to 18 years
* Recent (<6months) upper digestive endoscopy
* Ability to consent to participate in the study

Exclusion Criteria:

* Documented allergy to any of the available drugs
* Contraindications to any of the available drugs
* Antibiotics use for the last 4 weeks
* Previous gastric cancer
* Previous gastric surgery
* Pregnancy
* Breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | Approximately 1 month after treatment
  Confirmation of H. pylori eradication

CONTACTS AND LOCATIONS:
Locations (1):
- Vítor Bruno Macedo da Silva, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: Undecided